CLINICAL TRIAL: NCT06696391
Title: Venous Excess Ultrasound (VEXUS)-Guided Management Versus Usual Care in Patients with Septic Shock: a Pilot Randomized Controlled Trial
Brief Title: Venous Excess Ultrasound for Personalized Resuscitation in Septic Shock
Acronym: VESPER
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: London Health Sciences Centre (Other)
Responsible Party: Principal Investigator, John Basmaji, Critical Care Physician, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 125708
Record Dates: First submitted 2024-11-14; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-10

CONDITIONS: Septic Shock; Sepsis; Shock; Critical Care, Intensive Care; Resuscitation
Keywords: Randomized Controlled Trial; Ultrasound; Venous Congestion; Septic Shock; Pilot Study; Resuscitation
MeSH Terms: conditions — Shock, Septic; Sepsis; Shock; Hyperemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Venous Excess Ultrasound (VEXUS)-Guided Management (Experimental)
  Interventions: Other: Venous Excess Ultrasound (VEXUS)-Guided Management
- Control Arm (No Intervention): Investigators will provide patients with the standard of care according to the Surviving Sepsis Campaign guidelines. This includes fluid resuscitation, the recommended mean arterial pressure target of ≥65 mmHg, early broad-spectrum antibiotics, source control when applicable, vasopressor support with norepinephrine as the first-line agent, stress-dose corticosteroids, early nutrition, and lung-protective mechanical ventilation when required. Clinicians may utilize hemodynamics assessment tools such as dynamic measures of fluid responsiveness and point-of-care ultrasound.

INTERVENTIONS:
Other: Venous Excess Ultrasound (VEXUS)-Guided Management — Expert operators will perform VEXUS within 6 hours of randomization and repeat the assessment every 24 hours for 3 days, or until ICU discharge or death. After each assessment, investigators will grade the severity of venous congestion using a modified version of the VEXUS score and provide updated management recommendations.
  Patients without congestion will receive standard fluid management. For mild congestion, investigators will implement fluid restriction (e.g., minimizing maintenance fluids) while maintaining nutrition and blood product administration as clinically indicated. For moderate to severe congestion, investigators will 1. target negative fluid balance (-1 to -2L/24h) through fluid restriction and diuretics, 2. perform cardiac ultrasound to guide inotrope administration and optimize RV physiology, and 3. optimize PEEP for ventilated patients.
  All patients will receive the standard of care based on Surviving Sepsis Campaign guidelines.
  Arms: Venous Excess Ultrasound (VEXUS)-Guided Management

SUMMARY:
The goal of this pilot clinical trial is to determine if conducting a larger study using venous excess ultrasound (VEXUS) to guide fluid management in patients with septic shock is feasible. Septic shock is a life-threatening condition where infection causes dangerously low blood pressure. While fluids are essential for treatment, too much fluid can harm the kidneys and result in the need for dialysis. The main questions it aims to answer are:

1. Is it feasible to recruit patients, obtain consent, and follow the VEXUS-guided management protocol?
2. Does VEXUS-guided management, compared with usual care, improve the health and well-being of patients with septic shock?

Researchers will compare two groups: one receiving VEXUS-guided fluid management versus another receiving standard care, to assess the feasibility of a larger trial and explore whether VEXUS prevents fluid overload and kidney problems.

Participants in the VEXUS group will:

1. Undergo VEXUS scans every 24 hours for 3 days
2. Receive fluid management guided by VEXUS findings (including fluid restriction or removal if we identify venous congestion) and undergo cardiac ultrasound if we identify moderate to severe congestion
3. Be monitored for 28 days to track kidney function, need for dialysis, and survival.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥18 years)
2. Within 12 hours of meeting septic shock diagnosis based on following Sepsis-3 criteria: requirement for vasopressors to maintain organ perfusion, lactate > 2 mmol/L, and suspected or confirmed infection)
3. Within 48 hours of intensive care unit admission.

Exclusion Criteria:

1. Already receiving renal replacement therapy
2. Patients for whom a decision to initiate renal replacement therapy has been made prior to study enrolment
3. Patients who have limitations on medical therapy or restrictions on goals of care
4. Active bleeding causing hemodynamic instability
5. Veno-venous or veno-arterial extracorporeal membrane oxygenation
6. Previously enrolment in study
7. 10% or more of body surface area acute burn injury
8. Suspected or confirmed liver cirrhosis
9. Established allergy to sulfa drugs;
10. Patients receiving treatments that require continuous IV fluid infusions (e.g., diabetic ketoacidosis, diabetes insipidus)
11. Unable to measure fluid balance accurately
12. Contra-indication to study recommended interventions (e.g., diuretics, inotropes)
13. Unable to perform VEXUS due to anatomical barriers (e.g., surgical dressings);
14. Unable to complete VEXUS scan during the 6-hour resuscitation window
15. Moderate to Severe Tricuspid Regurgitation
16. Untreated Metabolic/biochemical findings (Hypokalemia [K+]< 3.0 mmol/L; metabolic alkalosis [Bicarbonate > 40 mmol/L and/or pH > 7.55], Hypomagnesemia [Mg2+] < 0.6, and Hypernatremia [Na+] > 155 mmol/L)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2027-12-28 (Estimated); Study Completion 2027-12-28 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | Up to 160 weeks
  Number of participants enrolled during the recruitment period who successfully complete study procedures and follow-up.

SECONDARY OUTCOMES:
Consent rate | From enrollment to the end of the study period at 28 days
  The total number of eligible participants consented divided by the total number of eligible participants approached for consent.
VEXUS scan completion rate | From enrollment to the end of treatment period at 3 days
  The number of participants who successfully undergo a VEXUS scan and, if applicable, cardiac evaluation, divided by the total number of participants randomized to the intervention arm.
Protocol Adherence | From enrollment to the end of treatment period at 3 days
  Intervention arm: For fluid balance adherence, we will calculate the proportion of participants who achieved the protocol-specified fluid balance targets on days 1 to 3, divided by the total number of participants in the intervention arm. This metric will account for participants who withdraw or deviate from the protocol. To assess adherence to inotrope initiation based on POCUS findings, we will determine the percentage of participants who received inotropes when indicated by POCUS results, as per protocol guidelines, divided by the total number of participants with POCUS findings warranting inotrope initiation.
  Control arm: The number of participants in the control arm who do NOT receive a VEXUS scan during the 28-day study period (or until ICU discharge or death) divided by the total number randomized to this arm.

OTHER OUTCOMES:
Adverse events | From enrollment to the end of treatment period at 3 days
  Metabolic abnormalities: hypokalemia < 3.0 mmol/L; hyponatremia <130 mmol/L, or hypernatremia > 155 mmol/L, metabolic alkalosis pH>7.55 or bicarbonate >40 mmol/L, and hypomagnesemia < 0.6 mmol/L) Hemodynamic events: hypotension episodes (defined as mean arterial pressure < 60 mmHg for 5 minutes or more), hypotension episodes requiring intervention (greater than 20% increase in vasopressor requirements from baseline or need for fluid bolus), tachyarrhythmias Organ Injury: acute kidney injury
  All adverse events will be reported daily for days 1 to 3
28-Day Mortality | From enrollment to 28 days
90-Day Mortality | From enrollment to 90 days
Duration of Vasoactive Medication | From enrollment to the discontinuation of vasoactive medication, assessed up to 52 weeks
  Defined as the time from initiation to the first successful discontinuation of vasopressors and inotropes, where successful discontinuation means no reinitiation for at least 12 consecutive hours
Days alive and free of vasoactive medications at 28 days | From enrollment to 28 days
Duration of mechanical ventilation | From enrollment to the discontinuation of mechanical ventilation, assessed up to 52 weeks
  Defined as the time from initiation to the first successful liberation of mechanical ventilation, where successful liberation means no reinitiation of mechanical ventilation for at least 12 consecutive hours
Days alive and free of mechanical ventilation at 28 days | From enrollment to 28 days
Need for Renal Replacement Therapy | From enrollment to 28 days
  Proportion of patients who require renal replacement therapy at 28 days
Days alive and free of renal replacement therapy at 28 days | From enrollment to 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Center, London, Ontario, Canada